CLINICAL TRIAL: NCT03328702
Title: Utilization of Continuous Positive Airway Pressure to Improve Swallow Function in Patients Post Total Laryngectomy
Brief Title: CPAP to Improve Swallow Function Post Total Laryngectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 908521
Record Dates: First submitted 2017-10-29; First posted 2017-11-01 (Actual); Results first posted 2024-12-24 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-12

CONDITIONS: Oropharyngeal Dysphagia; Laryngectomy; Status
Keywords: Dysphagia; Oropharyngeal dysphagia; Total Laryngectomy; Video Fluoroscopic Swallowing Exam (VFSE)
MeSH Terms: conditions — Deglutition Disorders | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Continue Positive Airway Pressure (Experimental): Continue Positive Airway Pressure during VFSE
  Interventions: Device: Continuous Positive Airway Pressure

INTERVENTIONS:
Device: Continuous Positive Airway Pressure — Apex XT Fit CPAP Machine

SUMMARY:
Investigator initiated prospective study to determine whether use of Continuous Positive Airway Pressure (CPAP) can improve the swallow function in patients who underwent total laryngectomy and are experiencing difficulty swallowing

DETAILED DESCRIPTION:
Total laryngectomy is a procedure that involves surgical removal of the larynx and separation of the digestive and airway tracts. The procedure is typically conducted for cases of laryngeal cancer and intractable aspiration. Following this procedure, patients are no longer at risk for aspiration; however some patients continue to experience difficulties in propulsion of food or drink throughout the pharynx. Previous research has demonstrated a reduction in pharyngeal contractile pressure and increased pharyngeal transit time in patients post laryngectomy. Continuous Positive Airway Pressure (CPAP) may assist bolus propulsion in these patients by increasing pressure in the direction of bolus flow. This study aims to evaluate the utility of a CPAP mask to improve pharyngeal swallow outcomes during Video Fluoroscopic Swallowing Exam (VFSE) in patients with dysphagia following total laryngectomy. This specific population could be well-suited for this application, since the digestive tract and airway are completely separate and there is no risk of the aspiration into the airway.

ELIGIBILITY:
Inclusion Criteria:

* Patients at least 2 months after total laryngectomy
* Undergoing Video Fluoroscopic Swallowing Examination

Exclusion Criteria:

* Patients with 100% neopharyngeal stenosis
* Patients with active cancer within 2 months of the study
* Patients with pharyngocutaneous fistula
* Vulnerable population: Adults unable to consent, Pregnant women, and Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2016-06-27 (Actual); Primary Completion 2022-11-08 (Actual); Study Completion 2022-11-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- UC Davis Medical Center, Sacramento, California, United States

REFERENCES:
- See also: Learn more or sign up for the study here! — https://studypages.com/s/a-study-of-continuous-positive-airway-pressure-cpap-to-improve-swallow-function-after-total-laryngectomy-784332/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Continue Positive Airway Pressure
Started | 4
Completed | 4
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Continue Positive Airway Pressure
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 56 (2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 4
Region of Enrollment [Number; unit: participants]
  United States | 4
Total Pharyngeal Transit Time @ Baseline (No CPAP) [Mean (Standard Deviation); unit: seconds] | 26.88 (12.5)

OUTCOME MEASURES:

1. Primary Outcome: Total Pharyngeal Transit Time (With CPAP)
Description: This is the time in seconds that it takes for a bolus to move from the oral cavity, through the pharynx, and into the so. It is measured in seconds and is the primary outcome measure.
Time Frame: During VFSE (1 day)
Population: The total pharyngeal transit time
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Continue Positive Airway Pressure
Number analyzed (Participants) | 4
seconds | 10.18 (8.5)
Statistical Analysis 1: Comparison: Continue Positive Airway Pressure; The null hypothesis is that there is no difference in total pharyngeal transit time with the use of CPAP; Test type: Superiority — Repeated measures ANOVA; p < 0.05, ANOVA — Repeated measures ANOVA, N=4; Repeated measures ANOVA; Mean Difference (Net) = 0.01

ADVERSE EVENTS:
Time Frame: 20 minutes (the approximate duration of the fluoroscopic swallow study).
Description: There were no adverse events
Arm/Group | Continue Positive Airway Pressure
All-Cause Mortality (participants affected / at risk) | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-05-20): https://cdn.clinicaltrials.gov/large-docs/02/NCT03328702/Prot_SAP_000.pdf